CLINICAL TRIAL: NCT00558168
Title: Electronic Study for Anastrozole Pharmacovigilance Evaluation
Acronym: E-SAFE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: ARI-IPEP-0104
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Early Breast Cancer
Keywords: Anastrazole; safety; early breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Collecting information regarding adverse events from patients on treatment with anastrazole with early stage breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal Early Invasive Breast Cancer Patients who are under anastrazole treatment, who have normal renal and hepatic functions.

Exclusion Criteria:

* Metastatic breast cancer patients, previous hormonal therapy, other malignancies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1850 (Actual)
Dates: Start 2004-01; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nejdet Uskent, Principal Investigator — Kadir Has University Medical School